CLINICAL TRIAL: NCT01711333
Title: A Multicenter, Therapeutic Used Study to Evaluate the Efficacy and Safety of Pletaal SR Capsule (Cilostazol) in Subjects With Peripheral Arterial Disease Symptom Due to Chronic Occlusive Arterial Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Pletaal SR Capsule (Cilostazol) in Subjects With Peripheral Arterial Disease Symptom Due to Chronic Occlusive Arterial Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 021-KOA-1102i
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Chronic Occlusive Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pletaal SR capsule (Experimental)
  Interventions: Drug: Pletaal SR capsule

INTERVENTIONS:
Drug: Pletaal SR capsule — two capsules once a day of Pletaal SR 100mg Capsules

SUMMARY:
This study is to evaluate symptomatic changes and safety before and after the administration of Pletaal® SR Capsules based on Peripheral Artery Questionnaire (PAQ) in subjects with peripheral arterial disease symptom due to chronic occlusive arterial disease (COAD).

DETAILED DESCRIPTION:
This is a multinational, single-arm, therapeutic used clinical trial. After screening in subjects with peripheral arterial disease symptom due to chronic occlusive arterial disease, the eligible subjects will be enrolled, followed by the administration of the study drug (two capsules qd of Pletaal SR 100mg Capsules) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female outpatients between 40 and 75 years of age,
2. Patients confirmed to have symptoms of peripheral arterial disease (including intermittent claudication, pain, coldness and fatigue) in the lower extremities,
3. Patients who have a steady symptom without significant improvement within 12 weeks prior to screening visit and whose PAQ score of the question number 3 is 3 or less at enrollment visit,
4. Ankle Branchial Index (ABI) ≤0.90 when measuring the pressure in a supine position after resting for 10 minutes,
5. Patients who are equal to or less than 10% of the difference in PAQ summary scores at between screening and enrollment,
6. Patients who have been fully explained about this study, voluntarily decided to participate in this study, and provided written informed consent.

Exclusion Criteria:

1. Patients with ischemic pain at rest or having ischemic ulcer or gangrene,
2. Patients with Ankle Branchial Index (ABI) ≤ 0.40
3. Patients who underwent sympathectomy or lower extremity arterial reparative surgery including endovascular procedures within 12 weeks prior to screening visit,
4. Patients diagnosed of deep vein thrombosis within 12 weeks prior to screening visit, (provided that patients with isolated calf vein thrombosis may be enrolled)
5. Patients with the following disease:

   * Patients who is on or needs the treatment for Congestive heart failure
   * Myocardial infarction which occurred within 24 weeks prior to screening visit
   * Patients who is on or needs the treatment for unstable angina pectoris,
6. Patients with hemorrhage (hemophilia, capillary fragility, intracranial hemorrhage, upper gastrointestinal hemorrhage, urinary hemorrhage, hemoptysis, vitreous hemorrhage, etc.) and predisposition to hemorrhage (active peptic ulcer, hemorrhagic stroke within the recent 24 weeks, suspected hemorrhage when administering cilostazol for wound due to surgery within the recent 12 weeks, and proliferative diabetic retinopathy),
7. PT, aPTT level greater than 1.5 times the upper limit of normal at screening visit,
8. Uncontrolled hypertension defined as ≥ 160 mmHg of systolic blood pressure or ≥ 100 mmHg of diastolic blood pressure,
9. Creatinine clearance(Ccr)a ≤ 25mL/min at screening a. Creatinine clearance (Ccr) is calculated by the following modified Cockcroft-Gault formula using the serum creatinine as determined by the site laboratory.

Ccr(mL/min)=[260-age(year)] x Body weight(kg) / 160 x Serum creatinine(mg/dL) (male) Ccr(mL/min)=[236-age(year)] x Body weight(kg) / 180 x Serum creatinine(mg/dL) (female), 10) AST or ALT level greater than 3 times the upper limit of normal at screening, 11) Total bilirubin level greater than 2 times the upper limit of normal at screening, 12) Type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus (HbA1c greater than 9%), 13) Patients determined ineligible to participate in this clinical trial at the discretion of Investigator due to critical diabetic complications (diabetic foot ulcer, foot deformity, etc.), 14) Female patients whose serum pregnancy test at screening or urine pregnancy test at enrollment is positive in case of childbearing potential and breastfeeding women,

* For female patients, those who have been at their postmenopause at least for one year or longer, who have no potential to be pregnant by surgery or procedure, or who agreed to use acceptable contraceptive methods (intrauterine device [loop or Mirena], double barrier method [diaphragm or condom/femidom + spermicide], vasectomy in spouse, oral contraceptives or non-oral contraceptives) throughout the entire study period,Female patients whose pregnancy test at screening is positive in case of childbearing potential or breastfeeding women 15) History of malignant disease (excluding treated basal cell or squamous cell carcinoma of skin) within 5 years prior to Screening. Resolution of a prior malignancy more than 5 years prior to Screening must be deemed as cured by the investigator, 16) Patients who have history of taking or plan to take the following medications:
* Cilostazol-containing medications within 12 weeks prior to screening visit,
* Antiplatelets (such as aspirin and ticlopidine), anticoagulants (such as warfarin), thrombolytics (such as urokinase and alteplase), prostaglandin E1 and its derivatives (such as alprostadil and limaprost), pentoxyfylline, beraprost, sarpogrelate and statin within 4 weeks prior to screening visit. However, aspirin (≤ 100 mg) or statin being taken for more than 4 weeks prior to screening visit may be administered at the same dose.
* Nitrates, papaverine, isoxsuprine, and NSAIDs within 4 weeks prior to screening visit. However, NSAIDs being taken for more than 4 weeks prior to screening visit may be administered at the same dose, 17) Patients with a history of hypersensitivity to cilostazol, 18) Patients who have received an investigational product or biological agent within 12 weeks prior to screening visit, 19) Patients who plans to enroll in another clinical trial (excluding observational studies) during this study, 20) Patients who needs to stop the Investigational Product because of scheduled operation, extraction of tooth or endoscopy, 21) Patients who are otherwise judged by the investigator to be inappropriate for inclusion in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-10-26 (Actual); Primary Completion 2014-05-20 (Actual); Study Completion 2014-08-18 (Actual)

PRIMARY OUTCOMES:
Summary score based on PAQ (Peripheral artery questionnaire) | Change from Baseline in PAQ summary score at Week 12

SECONDARY OUTCOMES:
Score of domain (physical limitation) based on PAQ | Change from Baseline in PAQ domain (physical limitation) at Week 12
Assessement based on HAQ-DI | Change from Baseline in HAQ-DI at Week 12
Score of domain(symptom) based on PAQ | Change from Baseline in PAQ domain(symptom) at Week 12
Score of domain(symptom stability) based on PAQ | Change from Baseline in PAQ domain(symptom stability) at Week 12
Score ofdomain(social limitation) based on PAQ | Change from Baseline in PAQ domain (social limitation) at Week 12
Score of domain(treatment satisfaction) based on PAQ | Change from Baseline in PAQ domain (treatment satisfaction) at Week 12
Score of domain(quality of life) based on PAQ | Change from Baseline in PAQ domain (quality of life) at Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- KYUNG-HEE UNIVERSITY HOSPITAL at GANGDONG, Seoul, South Korea